CLINICAL TRIAL: NCT03731013
Title: Mediterranean Diet and Physical Activity: is the Whole Better Than the Sum of Each Part ? Clinical and Mechanistic Perspectives
Brief Title: Combining a Mediterranean Diet With Physical Activity to Address Cardiometabolic Risk
Acronym: MEx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Benoit Lamarche, Study director, Laval University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: INAF-MEx 21628
Record Dates: First submitted 2018-10-22; First posted 2018-11-06 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Cardiometabolic Risk
MeSH Terms: interventions — Diet, Mediterranean; Exercise

STUDY DESIGN:
Intervention Model Description: Parallel group 2x2 factorial design clinical trial according to which participants will be randomly assigned to one of four 16-week intervention groups: 1- Mediterranean Diet alone; 2- Physical Activity alone ; 3- Combination of Mediterranean Diet and Physical Activity; 4- Control Group (no intervention).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Mediterranean diet (MedDiet) (Experimental)
  Interventions: Behavioral: Mediterranean diet (MedDiet)
- Physical activity (PA) (Experimental)
  Interventions: Behavioral: Physical activity (PA)
- Mediterranean diet and physical activity (Experimental)
  Interventions: Behavioral: Mediterranean diet and physical activity
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Mediterranean diet (MedDiet) — Participants randomized in the Mediterranean diet group without physical activity will be instructed and supported towards adhering to principles of the Mediterranean diet, without changes in physical activity habits.
  Arms: Mediterranean diet (MedDiet)
Behavioral: Physical activity (PA) — Participants randomized in the group physical activity without Mediterranean diet will participate in a structured, supervised PA program to achieve 150 min of moderate PA per week, without changes in dietary habits.
  Arms: Physical activity (PA)
Behavioral: Mediterranean diet and physical activity — The combination group (MedDiet + PA) will receive the combination of both interventions.
  Arms: Mediterranean diet and physical activity

SUMMARY:
There is little doubt scientifically that healthy eating, such as adhering to the Mediterranean diet (MedDiet) principles, is key for the prevention of cardiovascular disease (CVD). There is also convincing evidence for a strong inverse relationship between moderate intensity physical activity (PA) and mortality. Surprisingly, no study has yet formally documented how the combination of a MedDiet and regular PA improves cardiometabolic health in high-risk individuals. Why is this an important issue to address? On the one hand, a rigorous demonstration that the combination of a healthy diet and PA is better than the sum of each part in terms of cardiometabolic benefits will underpin the importance of advocating the combination of both modalities systematically to maximize health effects. Alternatively (and provocatively), results showing that healthy eating and PA have non-additive or non-synergistic effects will imply that one needs to adhere to only one of these two lifestyle modalities to maximizes cardiometabolic benefits. The overarching aim of this research is to test the hypothesis that consumption of a MedDiet combined with PA do act synergistically to improve cardiometabolic risk. The investigators hypothesize that healthy eating and PA act in synergy to reduce postprandial lipemia, a powerful independent risk factor for coronary heart disease.

DETAILED DESCRIPTION:
This is a randomized study with a 2X2 experimental factorial design. A total of 200 men and women recruited in the Quebec City area via various media will participate in this study. Eligible participants will be randomly assigned to one of four 16-week intervention groups: 1- Mediterranean Diet (MedDiet); 2- Physical Activity (PA); 3- Combination of MedDiet and PA; 4- Control Group. Depending on the group, the intervention involves support for nutritional and PA components at different times, in groups or individually. The subjects assigned to the MedDiet will receive certain foods each week to enhance adherence to the diet. Subjects assigned to the PA groups will have the opportunity to have one to two practices supervised by week by a team kinesiologist. All participants will have questionnaires to complete at different times during the study. These questionnaires will document several important aspects of the study including participants' health status, eating behaviours, hunger and satiety levels, eating and PA habits, motivation levels and well-being. Participants' diets will be assessed using a validated web 24-hour recall (R24W), which evaluates the food and beverages consumed during the 24 hours prior to the day they complete the questionnaire. This questionnaire will be completed over three randomly selected days on five occasions during the study. The level of PA will be evaluated using an accelerometer that objectively calculates energy expenditure. This device will be worn by participants for consecutive periods of 7 days, 5 times during the study.

Serum triglycerides (TG) concentrations after an oral fat load (35g of fat/m2 of body surface) and other the outcome variables will be measured in each group at baseline and at the end of the 16-week intervention. Specially, the fat load test will occur 2 days after the end of the intervention (114 days), so that the effect of the last exercise training bout has washed out. Cardiometabolic risk factors in the fasting state will be measured at baseline as well as twice at the end of the intervention, i.e. at 16 weeks (112 days) and at 16.3 weeks (114 days). The cardiorespiratory condition of the subjects will be evaluated during an maximal exercise test at the beginning and end of the 16-week intervention (112 days). Body composition will be assessed at the beginning and end of the intervention (112 days) by Dual Energy X-ray Absorptiometry (DEXA). Cardiac structure and function will be measured at the beginning and end (112 days) of the intervention using advanced echocardiographic imaging. Exercise capacity (VO2max) will measured by a modified Bruce protocol at the beginning and end (112 days) of the intervention. Fecal sample will be collected as an optional part of the study at baseline as well as at the end of the intervention (112 days). Deep 16S rDNA metagenomic analysis (in feces) as well as analyses of microbiota metabolites and endogenous bioactive lipid mediators in plasma will be used as surrogates of gut microbiota composition and function.

The primary objective is to compare the impact of each intervention and hence the potential synergistic impact of the MedDiet and PA on postprandial TG concentrations measured 4 hours after consumption of the oral fat load.

Secondary objectives are to compare the impact of each intervention and hence the potential synergistic impact of the MedDiet and PA on fasting concentrations of the following cardiometabolic risk factors: LDL-C, HDL-C, TG, CRP, adiponectin, IL-6, IL-8, TNFA-alpha, SBP, DBP. These comparisons will be performed on two sets of measures at the end of the intervention, i.e. at 16 week (112 days) and 2 days later (16.3 weeks, or 114 days). Secondary objectives also include the comparison of each intervention and hence the potential synergistic impact of the MedDiet and PA on cardiac structure and function and on exercise capacity (VO2max) measured at the end of the 16-week intervention (112 days).

Other pre-specified outcomes include assessment of the associations between changes in study outcomes and in abdominal fat levels as well as exploratory analyses of how the microbiota markers explain the difference between groups in cardiometabolic risk (exploratory objective).

ELIGIBILITY:
Inclusion Criteria:

* Waist circumference of 80 cm and over for women and 94 cm and over for men
* Serum triglyceride concentration of 1.5 mmol/L or higher
* For pre-menopausal women: regular cycle for at least 3 months, do not become pregnant or breastfeed
* For menopausal women: no hormone or stable dose for at least 6 months

Exclusion Criteria:

* Have a calculated Mediterranean score > 25
* Do > 100 minutes of moderate physical activity per week
* Weight change of > 5 kg in the last 3 months
* Presence of familial hypercholesterolemia, diabetes, history of CVD
* Take medications that affect inflammation and blood lipids
* Have taken anti-diabetic agents in the last 6 months
* Smoker
* Alcohol consumption >14 drinks per week
* Have allergies or aversions to components of the Mediterranean diet
* Follow a structured training program
* Dieting or having a special diet
* Inability to engage in a physical activity program

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2018-10-22 (Actual); Primary Completion 2023-04-24 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
1. Serum 4-hour post-prandial TG concentrations | 16.3 week (114 days)
  Serum TG concentrations (mmol/l) will be measured 4 hours after ingestion of a fatty meal (fat load), at the end of the 16-week intervention in all subjects in each group. The fat load will be conducted 48 hours after the last exercise training session in the PA groups (hence at 16.2 weeks, or 114 days). Analyses will be adjusted for 4-hr postprandial TG values measured at baseline.

SECONDARY OUTCOMES:
Serum fasting TG concentrations | 16 week (112 days)
  Fasting serum TG concentrations (mmol/l) will be measured at the end of the 16-wk intervention in all subjects in each group. Analyses will be adjusted for fasting TG values measured at baseline.
Serum fasting TG concentrations | 16.3 week (114 days)
  Fasting serum TG concentrations (mmol/l) will be measured 2 days after the end of the 16-wk intervention in all subjects in each group (hence 16.3 weeks, or 114 days). Analyses will be adjusted for fasting TG values measured at baseline.
Serum fasting LDL-C concentrations | 16 week (112 days)
  Fasting serum LDL-C concentrations (mmol/l) will be measured at the end of the 16-wk intervention in all subjects in each group. Analyses will be adjusted for fasting LDL-C values measured at baseline.
Serum fasting LDL-C concentrations | 16.3 week (114 days)
  Fasting serum LDL-C concentrations (mmol/l) will be measured 2 days after the end of the 16-wk intervention in all subjects in each group (hence 16.3 weeks, or 114 days). Analyses will be adjusted for fasting LDL-C values measured at baseline.
Serum fasting HDL-C concentrations | 16 week (112 days)
  Fasting serum HDL-C concentrations (mmol/l) will be measured at the end of the 16-wk intervention in all subjects in each group. Analyses will be adjusted for fasting HDL-C values measured at baseline.
Serum fasting HDL-C concentrations | 16.3 week (114 days)
  Fasting serum HDL-C concentrations (mmol/l) will be measured 2 days after the end of the 16-wk intervention in all subjects in each group (hence 16.3 weeks, or 114 days). Analyses will be adjusted for fasting HDL-C values measured at baseline.
Serum fasting CRP concentrations | 16 week (112 days)
  Fasting serum CRP concentrations (mg/ l) will be measured at the end of the 16-wk intervention in all subjects in each group. Analyses will be adjusted for fasting CRP values measured at baseline.
Serum fasting CRP concentrations | 16.3 week (114 days)
  Fasting serum CRP concentrations (mg/ l) will be measured 2 days after the end of the 16-wk intervention in all subjects in each group (hence 16.3 weeks, or 114 days). Analyses will be adjusted for fasting CRP values measured at baseline.
Serum fasting adiponectin concentrations | 16 week (112 days)
  Fasting serum adiponectin concentrations (mg/l) will be measured at the end of the 16-wk intervention in all subjects in each group. Analyses will be adjusted for fasting adiponectin values measured at baseline.
Serum fasting adiponectin concentrations | 16.3 week (114 days)
  Fasting serum adiponectin concentrations (mg/l) will be measured 2 days after the end of the 16-wk intervention in all subjects in each group (hence 16.3 weeks, or 114 days). Analyses will be adjusted for fasting adiponectin values measured at baseline.
Serum fasting IL-6 concentrations | 16 week (112 days)
  Fasting serum IL-6 concentrations (pmol/l) will be measured at the end of the 16-wk intervention in all subjects in each group. Analyses will be adjusted for fasting IL-6 values measured at baseline.
Serum fasting IL-6 concentrations | 16.3 week (114 days)
  Fasting serum IL-6 concentrations (pmol/l) will be measured 2 days after the end of the 16-wk intervention in all subjects in each group (hence 16.3 weeks, or 114 days). Analyses will be adjusted for fasting IL-6 values measured at baseline.
Serum fasting IL-18 concentrations | 16 week (112 days)
  Fasting serum IL-18 concentrations (pmol/l) will be measured at the end of the 16-wk intervention in all subjects in each group. Analyses will be adjusted for fasting IL-18 values measured at baseline.
Serum fasting IL-18 concentrations | 16.3 week (114 days)
  Fasting serum IL-18 concentrations (pmol/l) will be measured 2 days after the end of the 16-wk intervention in all subjects in each group (hence 16.3 weeks, or 114 days). Analyses will be adjusted for fasting IL-18 values measured at baseline.
Serum fasting TNF-alpha concentrations | 16 week (112 days)
  Fasting serum TNF-alpha concentrations (pmol/l) will be measured at the end of the 16-wk intervention in all subjects in each group. Analyses will be adjusted for fasting TNF-alpha values measured at baseline.
Serum fasting TNF-alpha concentrations | 16.3 week (114 days)
  Fasting serum TNF-alpha concentrations (pmol/l) will be measured 2 days after the end of the 16-wk intervention in all subjects in each group (hence 16.3 weeks, or 114 days). Analyses will be adjusted for fasting TNF-alpha values measured at baseline.
Systolic blood pressure (SBP) | 16 week (112 days)
  SBP (mmHg) will be measured at the end of the 16-wk intervention in all subjects in each group. Analyses will be adjusted for SBP values measured at baseline.
Systolic blood pressure (SBP) | 16.3 week (114 days)
  SBP (mmHg) will be measured 2 days after the end of the 16-wk intervention in all subjects in each group (hence 16.3 weeks, or 114 days). Analyses will be adjusted for SBP values measured at baseline.
Diastolic blood pressure (DBP) | 16 week (112 days)
  DBP (mmHg) will be measured at the end of the 16-wk intervention in all subjects in each group. Analyses will be adjusted for DBP values measured at baseline.
Diastolic blood pressure (DBP) | 16.3 week (114 days)
  DBP (mmHg) will be measured 2 days after the end of the 16-wk intervention in all subjects in each group (hence 16.3 weeks, or 114 days). Analyses will be adjusted for DBP values measured at baseline.
Maximal oxygen consumption (VO2max) | 16 week (112 days)
  Maximal oxygen consumption, a metric of cardiorespiratory fitness, will be measured by a modified Bruce protocol at the end of the 16-wk intervention in all subjects in each group. Analyses will be adjusted for VO2max values measured at baseline.
Left ventricular (LV) global longitudinal strain | 16 week (112 days)
  LV global longitudinal strain in % will be measured using transthoracic echocardiogram and speckle tracking for systolic and diastolic strain/strain rates. Analyses will be adjusted for LV global longitudinal strain values measured at baseline.
Right ventricular (RV) global longitudinal strain | 16 week (112 days)
  RV global longitudinal strain in % will be measured using transthoracic echocardiogram and speckle tracking for systolic and diastolic strain/strain rates. Analyses will be adjusted for RV global longitudinal strain values measured at baseline.
Cardiac chamber volumes | 16 week (112 days)
  Cardiac chamber volumes (cm3) will be measured using transthoracic echocardiogram with pulse-wave, continuous-wave and tissue Dopplers. Analyses will be adjusted for cardiac chamber volumes measured at baseline.

OTHER OUTCOMES:
Change (week 0 vs week 16) in android obesity | week 0 and week 16 (112 days)
  Levels of total and abdominal fat (volume in cm3) will be measured at baseline and post-intervention (16 week) by DEXA in all participants. Associations between changes in study outcomes and in body fat distribution will be assessed by correlational and multiple regression analyses
Gut microbiota | 16 week (112 days)
  These are exploratory analyses in a subset of participants only. Deep 16S rDNA metagenomic analysis (in feces) as well as analyses of microbiota metabolites and endogenous bioactive lipid mediators in plasma will be used as surrogates of gut microbiota composition and function in these exploratory analyses of between group differences. Analyses will be adjusted for baseline values.

CONTACTS AND LOCATIONS:
Overall Officials: Benoît Lamarche, PhD, Principal Investigator — Laval University
Locations (1):
- Institute of Nutrition and Funtional Foods, Québec, Canada